CLINICAL TRIAL: NCT01997372
Title: Different Doses of Anti-thymocyte Globin With 2.5 or 3.75mg/kg to Treat Child Severe Aplastic Anemia
Brief Title: Different Doses of Anti-thymocyte Globin to Treat Child Severe Aplastic Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiaofan Zhu, Department of Pediatrics, Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xzhu
Record Dates: First submitted 2012-03-01; First posted 2013-11-28 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Severe Aplastic Anemia
Keywords: ATG; SAA; immunosuppressive treatment; cyclosporine
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high dose ATG,low dose ATG (Experimental)
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: ATG — Drug ATG:2.5mg/kg/d or 3.75mg/kg/d for 5 days; Drug Cyclosporine A (CSA):3-10mg/kg/d ,Adjust the dose to maintain drug levels between 150 and 300ng/ml; Drug prednisone:1mg/kg/d,d1-21 from the first dosage of ATG; Drug Granulocyte Colony-Stimulating Factor(G-CSF):5ug/kg/d until absolute neutrophil count (ANC) >1×109/L.

SUMMARY:
Severe acquired aplastic anaemia (SAA) is a life-threatening disease characterized by pancytopenia and hypoplastic bone marrow. Immunosuppressive treatment with antithymocyte globulin (ATG)and cyclosporine remain the standard regimen with response rates of 70% or more and excellent overall survival. However ,there are no clinical trials to illustrate the response and complete remission rate with different doses of ATG.And there are no data reported on children with SAA so far.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of childhood acquired severe aplastic anemia(SAA)

Exclusion Criteria:

* clinical diagnosis of no childhood acquired severe aplastic anemia(SAA)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
the response and complete remission rate with different doses of ATG to treat child severe aplastic anemia | 1 years
  Complete response (CR) was defined as achieving normal levels of hemoglobin adjusted for age, platelet count >100×109/L, and ANC>1.5×109/L. Partial response (PR) was defined as transfusion independence, reticulocyte count >30×109/L, platelet count >20×109/L, and ANC >0.5×109/L above the baseline. Persistence of transfusion requirement or death was evidence of no response (NR).

SECONDARY OUTCOMES:
the relapse rate with different doses of ATG to treat child severe aplastic anemia | 4-10 years
  relapse was defined as transfusion dependence again; or progressed to paroxysmal nocturnal hemoglobinuria (PNH) /acute myeloid leukemia/myelodysplasia syndrome (MDS); or CSA dependence

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Result] Camitta BM, Rappeport JM, Parkman R, Nathan DG. Selection of patients for bone marrow transplantation in severe aplastic anemia. Blood. 1975 Mar;45(3):355-63. PMID 1090310